CLINICAL TRIAL: NCT02318784
Title: Phase II Study of Carfilzomib for the Treatment of Patients With Advanced Neuroendocrine Cancers
Brief Title: Carfilzomib for the Treatment of Patients With Advanced Neuroendocrine Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 195
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2022-06

CONDITIONS: Neuroendocrine Cancer
Keywords: neuroendocrine malignancies; pancreatic neuroendocrine tumors (PNETs); gastrointestinal (GI) carcinoids; carfilzomib; Kyprolis; proteasome inhibitors
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Carcinoid Tumor | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib (Experimental): Carfilzomib will be administered as intravenous (IV) infusion over 30 minutes on Days 1, 2, 8, 9, 15 and 16 of each 28-day cycle.
  Cycle 1: First two doses of Carfilzomib 20 mg/m2 IV; subsequent doses at 56 mg/m2 IV
  Cycle 2 onwards: Carfilzomib 56 mg/m2 IV
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib
  Other Names: Kyprolis

SUMMARY:
The purpose of this study is to determine if carfilzomib is safe and effective in the treatment of patients with advanced neuroendocrine tumors.

DETAILED DESCRIPTION:
Neuroendocrine malignancies such as pancreatic neuroendocrine tumors (PNETs) and gastrointestinal (GI) carcinoids, are generally rare but their incidences are increasing. In vitro and in vivo studies have shown that proteasome inhibitors have activity against a variety of tumor types. Carfilzomib (Kyprolis®) is an irreversible proteasome inhibitor with a favorable safety profile that has been studied in a variety of hematologic and solid tumors. Carfilzomib received accelerated approval from the U.S. FDA in 2012, based on a favorable response rate, for the treatment of patients with multiple myeloma who received at least two prior therapies, and demonstrated disease progression within 60 days of completing the last therapy. In this multi-center study, the investigators propose to evaluate carfilzomib for the treatment of patients with advanced neuroendocrine cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with biopsy-proven advanced, unresectable or metastatic, well-to-moderately differentiated (or low grade) neuroendocrine carcinoma, including typical carcinoid, pancreatic islet cell and other well-to-moderately differentiated neuroendocrine carcinomas.
2. Measurable disease per Response Evaluation Criteria in Solid Tumors RECIST v 1.1 criteria.
3. Patients currently receiving or previously treated with single agent sandostatin LAR® are eligible. However, this is not a mandatory criterion to be included in the study.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
5. Adequate hematologic, renal, and hepatic function.
6. Predicted life expectancy > 12 weeks.

Exclusion Criteria:

1. Patients with poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, globlet cell carcinoid, atypical carcinoid, anaplastic carcinoid, pulmonary neuroendocrine and small cell carcinoma are not eligible.
2. Patients who had radiation therapy, hormonal therapy, biologic therapy, investigational agents, or chemotherapy for cancer within 21 days or 5 half-lives of any chemotherapy or biologic/targeted agent, whichever is longer, prior to first treatment day of the study.
3. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would impair the ability of the patient to receive protocol treatment.
4. Major surgical procedures ≤28 days of beginning study drug, or minor surgical procedures ≤7 days. No waiting required following port-a-cath placement.
5. Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 2 weeks prior to study entry and there is no evidence of central nervous system disease progression, mild neurologic symptoms, and no requirement for chronic corticosteroid therapy.
6. Known diagnosis of human immunodeficiency virus, hepatitis B or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (10):
- United States (10):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Research Medical Center, Kansas City, Missouri
  - Oncology Hematology Care, INC., Cincinnati, Ohio
  - Spartanburg Regional Medical Center/Gibbs Cancer Center, Spartanburg, South Carolina
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Center for Cancer and Blood Disorders, Fort Worth, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Carfilzomib: Carfilzomib - administered as an intravenous (IV) infusion over 30 minutes on Days 1, 2, 8, 9, 15, and 16 of each 28-day cycle.
  Cycle 1: First two doses of Carfilzomib 20 mg/m^2 IV; subsequent doses at 56 mg/m2 IV
  Cycle 2 onwards: Carfilzomib 56 mg/m^2 IV
Period: Overall Study
Arm/Group | Carfilzomib
Started | 62
Completed | 0
Not Completed | 62
Not completed — Adverse Event | 13
Not completed — Death | 2
Not completed — Progressive Disease | 37
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Population: Full analysis set - all enrolled patients who receive at least one full or partial dose of the study group and who have measurable disease at baseline
Arm/Group | Carfilzomib
Number analyzed (Participants) | 62
Age, Continuous [Median (Full Range); unit: years] | 63 [28 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Percentage of participants with confirmed complete response (CR) or partial response (PR) (i.e. 2 CRs or PRs at least 4 weeks apart) to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1) CR=disappearance of all target lesions. PR=at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: every 3 cycles (1 cycle= 28 days) until treatment discontinuation up to 4 years
Population: All enrolled patients who received at least one full or partial dose of the study drug and who had measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 62
percentage of participants | 3.226 [0.4 to 11.2]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of participants with complete response (CR), partial response (PR), or stable disease (SD) (≥ 6 cycles) according to RECIST v1.1 criteria. Complete Response is defined per RECIST as the disappearance of all target/non-target lesions and normalization of tumor markers. Partial Response is defined per RECIST as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Stable disease is defined per RECIST as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest (nadir) sum LD since the treatment started.
Time Frame: every 3 cycles (1 cycle= 28 days) until treatment discontinuation up to 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 62
percentage of participants | 58 [44.8 to 70.5]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Measured from Day 1 of study drug administration to disease progression as defined by RECIST v1.1, or death on the study. Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or unequivocal progression of non-target lesions or the appearance of one or more new lesions. Patients who did not have disease progression or death documented were censored on the date of the last visit with adequate assessment.
Time Frame: up to 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib
Number analyzed (Participants) | 62
months | 8 [2.9 to 11.1]

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events as a Measure of Safety and Tolerability
Description: The number of treatment-emergent adverse events will be graded utilizing the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03
Time Frame: From the day of the first dose to 30 days after the last dose of study medication, up to 4 years
Population: All enrolled patients who received at least one full or partial dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 62
Participants | 56

ADVERSE EVENTS:
Time Frame: From the day of the first dose to 30 days after the last dose of study medication, up to 4 years
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were collected from the day of the first dose to 30 days after the last dose of the study medication and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Arm/Group | Carfilzomib
All-Cause Mortality (participants affected / at risk) | 10/62
Serious Adverse Events (participants affected / at risk) | 31/62
Other Adverse Events (participants affected / at risk) | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib (N=62)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Ectopic ACTH syndrome (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (8)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Malignant hypertension (Vascular disorders) | 1 (1)
Ticuspid valve replacement (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib (N=62)
Anaemia (Blood and lymphatic system disorders) | 12 (41)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (89)
Acute left ventricular failure (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Ear pruritus (Ear and labyrinth disorders) | 1 (1)
Ectopic ACTH syndrome (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 2 (3)
Diplopia (Eye disorders) | 1 (1)
Eye haematoma (Eye disorders) | 1 (1)
Eye swelling (Eye disorders) | 1 (2)
Lacrimation increased (Eye disorders) | 1 (1)
Periorbital oedema (Eye disorders) | 2 (4)
Vision blurred (Eye disorders) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 10 (15)
Abdominal pain (Gastrointestinal disorders) | 11 (19)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6)
Abdominal rigidity (Gastrointestinal disorders) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (15)
Defaecation urgency (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 26 (70)
Discoloured vomit (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Enteritis (Gastrointestinal disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 8 (10)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 37 (74)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1)
Pancreatic failure (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Retching (Gastrointestinal disorders) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 2 (3)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 32 (66)
Asthenia (General disorders) | 10 (14)
Catheter site bruise (General disorders) | 1 (1)
Catheter site inflammation (General disorders) | 1 (1)
Catheter site pain (General disorders) | 3 (3)
Catheter site related reaction (General disorders) | 2 (2)
Chest pain (General disorders) | 4 (4)
Chills (General disorders) | 12 (29)
Early satiety (General disorders) | 1 (1)
Fatigue (General disorders) | 33 (65)
Feeling hot (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (2)
Generalised oedema (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Infusion site pain (General disorders) | 1 (1)
Localised oedema (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 20 (33)
Pain (General disorders) | 7 (8)
Peripheral swelling (General disorders) | 4 (4)
Pyrexia (General disorders) | 18 (35)
Thirst (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 5 (7)
Chronic sinusitis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (2)
Ear infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (2)
Eye infection viral (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 3 (3)
Oral herpes (Infections and infestations) | 3 (3)
Perirectal abscess (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (4)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 8 (15)
Urinary tract infection (Infections and infestations) | 4 (12)
Wound infection (Infections and infestations) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (4)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase (Investigations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 6 (11)
Ammonia increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 6 (15)
Blood alkaline phosphatase increased (Investigations) | 6 (19)
Blood bilirubin increased (Investigations) | 6 (19)
Blood calcium increased (Investigations) | 1 (1)
Blood creatine increased (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 8 (22)
Blood glucose increased (Investigations) | 2 (3)
Blood potassium decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 2 (6)
Body temperature increased (Investigations) | 1 (2)
Brain natriuretic peptide increased (Investigations) | 1 (1)
Cardiac murmur (Investigations) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 2 (3)
Creatinine renal clearance increased (Investigations) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (5)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 9 (72)
Protein total decreased (Investigations) | 1 (1)
Respiratory rate increased (Investigations) | 1 (2)
Staphylococcus test positive (Investigations) | 1 (1)
Transferrin saturation decreased (Investigations) | 1 (1)
Urine bilirubin increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 9 (15)
Weight increased (Investigations) | 2 (2)
White blood cell count increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 12 (17)
Dehydration (Metabolism and nutrition disorders) | 10 (21)
Fluid retention (Metabolism and nutrition disorders) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (5)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (10)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 3 (3)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (21)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (9)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (5)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (9)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 14 (14)
Dysgeusia (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 26 (41)
Hypersomnia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3)
Lethargy (Nervous system disorders) | 2 (3)
Memory impairment (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 14 (21)
Irritability (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (4)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Chromaturia (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (7)
Dysuria (Renal and urinary disorders) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (21)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (26)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (4)
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 6 (7)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (6)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (3)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 4 (4)
Hot flush (Vascular disorders) | 4 (5)
Hypertension (Vascular disorders) | 16 (21)
Hypotension (Vascular disorders) | 7 (7)
Pallor (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT02318784/Prot_SAP_000.pdf